CLINICAL TRIAL: NCT02206568
Title: A Randomised Trial Investigating Pharmacokinetic Properties of Ultra-Rapid-Acting Insulin Lispro (URAL) in Subjects With Type 1 Diabetes Mellitus
Brief Title: Pharmacokinetics of Ultra-Rapid-Acting Insulin Lispro (URAL) in Type 1 Diabetes Mellitus
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Sponsor: Perosphere Pharmaceuticals Inc, a wholly owned subsidiary of AMAG Pharmaceuticals, Inc. (Industry)
Collaborators: Profil Institut für Stoffwechselforschung GmbH (Industry)
Responsible Party: Sponsor
Organization: AMAG Pharmaceuticals, Inc. (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: Triple | Purpose: Basic Science
Other Study IDs: PER511
Record Dates: First submitted 2014-07-30; First posted 2014-08-01 (Estimated); Last update posted 2020-07-15 (Actual); Status verified 2015-05

CONDITIONS: Type 1 Diabetes Mellitus
Keywords: diabetes mellitus; phase 1; insulin lispro; male subjects
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- URAL vs. Insulin lispro (Experimental): Each subject will randomly be allocated to a treatment sequence consisting of 2 dosing visits during which the subject in a euglycaemic clamp setting will receive either a single dose of insulin lispro or URAL at predefined fixed dose levels in a randomized order.
  Interventions: Drug: URAL

INTERVENTIONS:
Drug: URAL
  Other Names: Ultra-Rapid-Acting Insulin Lispro

SUMMARY:
To compare the early pharmacokinetic exposure of URAL and insulin lispro (ILisp).

DETAILED DESCRIPTION:
To compare the total pharmacodynamic response of URAL and insulin lispro.

To compare the total pharmacokinetic exposure between URAL and insulin lispro.

To assess the safety and tolerability of URAL and insulin lispro.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent
2. Male subjects age 18-65 years inclusive
3. Type 1 diabetes mellitus diagnosed clinically >= 12 months
4. Treatment with multiple daily insulin injections or CSII >= 12 months
5. Current total daily insulin treatment <1.2 (I)U/kg/day
6. Current total daily bolus insulin treatment <0.7 (I)U/kg/day
7. Body mass index 18.0-30.0 kg/m2 inclusive
8. HbA1c =<9.0% by local laboratory analysis (one retest within a week is permitted with the result of the last test being conclusive)
9. C-peptide =< 0.30 nmol/L

Exclusion Criteria:

1. Known or suspected hypersensitivity to trial products or related products
2. Previous participation in this trial. .
3. Receipt of any non-marketed investigational product within 3 months
4. Clinically significant abnormal haematology, biochemistry, liver enzymes, or coagulation screening tests
5. Suffer from or history of a life threatening disease or any clinically significant cardiovascular, respiratory, metabolic, renal, hepatic, gastrointestinal, endocrinological, haematological, dermatological, venereal , neurological, psychiatric diseases or other major disorders
6. History of deep leg vein thrombosis or a frequent appearance of deep leg vein thrombosis in 1st degree relatives
7. Cardiac problems defined as decompensated heart failure (New York Heart Association class III and IV) at any time and/or angina pectoris within the last 12 months and/or acute myocardial infarction at any time.
8. Supine blood pressure at screening outside the range of 90-140 mmHg for systolic or 50-90 mmHg for diastolic . Pulse outside 50 to 90 bpm.
9. Clinically significant abnormal ECG at screening.
10. Proliferative retinopathy or maculopathy and/or severe neuropathy, in particular autonomic neuropathy.
11. Any disease or condition that, in the opinion of the Investigator, would represent an unacceptable risk for the subject's safety.
12. Subject positive for HBs-Ag, HCV-Ab
13. Positive result to the screening test for HIV-1 antibodies, HIV-2 antibodies, or HIV-1 antigen according to locally used diagnostic testing.
14. History of multiple and/or severe allergies to drugs or foods or a history of severe anaphylactic reaction.
15. Subject who has donated blood or plasma in the past month or more than 500 mL within 3 months.
16. Surgery or trauma with significant blood loss (more than 500 mL) within 3 months.
17. Current treatment with systemic (oral, IV, or inhaled) corticosteroids, monoamine oxidase inhibitors, NSAID, prostaglandin blockers, systemic non-selective beta-blockers, growth hormone (last 3 months), non-routine vitamins or herbal products (last 2 weeks). Thyroid hormones are not allowed unless the use of these has been stable during the last 3 months. Routine vitamins are permitted up to 48 hours prior to dosing.
18. Significant history of alcoholism and/or drug/chemical abuse as per Investigator's judgement or a positive result in the urine drug/alcohol breath test screen at the screening visit.
19. Heavy smoker
20. Not able or willing to refrain from smoking and use of nicotine.
21. Recurrent severe hypoglycaemia (more than 1 severe hypoglycaemia event during the last 12 months) or hypoglycaemic unawareness.
22. Subject with mental incapacity or language barriers precluding adequate understanding.
23. Potentially non-compliant or uncooperative during the trial.
24. Any condition that would interfere with trial participation or evaluation of results.
25. No relevant lipodystrophy within the area of drug administration and Doppler sonography.

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-06; Primary Completion 2014-08 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics of URAL | 1 day
  Area under the serum insulin lispro concentration-time curve from 0-30 minutes after administration

SECONDARY OUTCOMES:
Onset of appearance of serum insulin lispro | 1 day
  Measurement of time to reach insulin lispro concentration >30 pmol/L in the serum
Number of subjects with adverse events | 1 day
  Assessment of safety and tolerability of URAL

CONTACTS AND LOCATIONS:
Overall Officials: Alin Stirban, MD, Principal Investigator — Profil Institut fur Stoffwechselforschung GmbH
Locations (1):
- Profil Institut fur Stoffwechselforschung GmbH, Neuss, Germany